CLINICAL TRIAL: NCT07394179
Title: Transforming Channel Shape Osteotomy Into Tunnel Shape Osteotomy for Zygomatic Implant. A Randomized Control Trial
Brief Title: Transforming Channel Osteotomy Into Tunnel Osteotomy in Zygomatic Implant Preparation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, haitham ahmed mohammed elmaergy, doctor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Grafting with zygoma implants
Record Dates: First submitted 2025-12-04; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Zygomatic Implants
Keywords: Zygomatic implants; Grafting; Tunnel and channel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): Zygomatic implants placed in Channel shape osteotomy with using xenogenic malleable bone shell to convert osteotomy type to tunnel osteotomy.
  Interventions: Procedure: Group A
- group B (Placebo Comparator): Zygomatic implants placed in Channel shape osteotomy with only soft tissue augmentation by using buccal bad of fat.
  Interventions: Procedure: Group B

INTERVENTIONS:
Procedure: Group A — after zygomatic implant placed with channel shape osteotomy,Wetting, trimming and fixation of xenogenic lamina shell buccal to placed zygomatic implants in combination with xenogenic particulate form to fill all gaps between lamina from one side and native bone and implant from other side
  Arms: group A
Procedure: Group B — after zygomatic implant placed with channel shape osteotomy ,Blunt dissection to buccal space to extract buccal pad of fat which will be mobilized and advanced to cover buccal surface of zygomatic implants and fixed over it with either suturing to palatal mucosa or with bone tacs
  Arms: group B

SUMMARY:
The evolution of zygomatic implant techniques, from the original procedures to the Zygomatic Anatomy-Guided Approach (ZAGA), has significantly improved outcomes for patients with severe maxillary atrophy. Despite these advancements, challenges such as peri-implant tissue recession, sinus complications, and aesthetic concerns persist. Bone augmentation and soft tissue enhancement techniques, including sinus lifts, connective tissue grafts, and buccal fat pad utilization, have been employed to address these issues with varying degrees of success. However, the need for predictable and stable bone regeneration and soft tissue contouring remains critical for long-term implant success.

The following study aims to assess bone gain, soft tissue contour, and stability after using bone lamina shell, providing a potential solution to enhance peri-implant tissue integrity and optimize functional and aesthetic outcomes in zygomatic implant rehabilitation

DETAILED DESCRIPTION:
The term "tunnel osteotomy" is used because the alveolar osseous entry point has a floor, lateral walls, and a more or less complete roof. When a tunnel osteotomy was chosen, the sinus membrane was perforated at the time of completion of the antrostomy. The objective was to achieve osseointegration at the neck level also to seal the sinus entrance in the long-term using: (1) a stable zygomatic implant with (2) a suitable threaded neck section (3) bordered by enough bone at the coronal entry, (4) stabilized by adequate apical zygomatic anchorage; and (5) connected to a rigid prosthesis that provides adequate masticatory load distribution. The "tunnel osteotomy" was also employed in ZAGA Type 3 cases when the alveolar bone adopts a triangular, buccally inclined, profile and the maxillary anterior wall was concave(23).

When inadequate residual bone architecture at the crestal level (less than 4 mm of thickness) was measured, the coronal osteotomy was buccally shifted to prevent future sinus or nasal-oral communication/fistula. Implant beds were designed to be carved as much as possible into both the buccal alveolar and maxillary wall bone with the limits of sinus lining integrity. This osteotomy type is known as a "channel osteotomy" and is noted when lateral walls and floor are present but with no roof(23).

On analyzing the evolution of the abovementioned technique (ZAGA), it is seen that the position of the neck of the zygomatic implants has been mobilized laterally from an intrasinus position to an extrasinus position. Different anterior techniques have thus sought to avoid maxillary sinus complications(19,24,25). However, hard and soft tissue infective and aesthetic complications (exposure of the implant threads) were detected(26-28).

Peri-implant hard and soft tissues are crucial for avoiding complications around conventional implants. Two aspects have been studied in this regard: buccal cortical bone and the thickness and width of the peri-implant keratinized mucosa. On the one hand, a recent systematic review has reported that a buccal cortical thickness of close to 2 mm was associated with less vertical bone resorption and less mucosal recession(29).

On the other hand, the presence of sufficient keratinized mucosa thickness exerts a protective effect against marginal bone loss(30,31). These abovementioned concepts to minimum necessary peri-implant tissues could be extrapolated to zygomatic implants. A number of techniques for bone and soft tissue enhancement around zygomatic implants have been described, with high success rates.

Regarding bone regeneration, a sinus lift during the zygomatic implant placement has been proposed (32). Regarding soft tissue enhancement, dissection of the buccal fat pad and the ZAGA "Scarf Graft" (pediculate connective tissue grafting [26]) have been utilized to prevent buccal mucosal recession(33). Chow et al. described a simultaneous sinus lift for reducing oroantral communications and subsequent maxillary sinus infections in zygomatic implants(34).

Hinze et al. with Chow's technique described an increase in peri-implant bone around the coronal part of the implant (buccal bone 1.4 ± 0.5 mm and palatal bone 4.3 ± 0.4 mm) at 6 months which same results of Peñarrocha et al study showed similar bone gained width(34,35).

Peri-implant bone defects or thin buccal/palatal corticals were regenerated with a mixture of particulate synthetic bone graft (beta-phosphate tricalcium (KeraOs ®, Keramat, Spain)) with autogenous bone and resorbable collagen membranes (Creos Xenoprotect ®, Nobel Biocare, Sweden) fixed with surgical pins (Meisinger ®, Sanhigia, Spain). Management of the soft tissue without flap pressure was achieved through two-plane suturing (horizontal double and simple stitches). Bone regeneration was performed palatal, buccal or palatal and buccal(35).

Palatal rotated connective tissue flaps or free connective tissue grafts were performed to improve buccal soft tissues around the zygomatic implants. Palatal rotated flaps were fixed buccally to the zygomatic implants using resorbable sutures through small perforations created in the bone alveolar crest mesial and distal of the zygomatic implant. Free connective tissue grafts were collected from the palatal flap and fixed buccally around the coronal part of the zygomatic implants by two surgical pins(35).

The evolution of zygomatic implant techniques, from the original procedures to the Zygomatic Anatomy-Guided Approach (ZAGA), has significantly improved outcomes for patients with severe maxillary atrophy. Despite these advancements, challenges such as peri-implant tissue recession, sinus complications, and aesthetic concerns persist. Bone augmentation and soft tissue enhancement techniques, including sinus lifts, connective tissue grafts, and buccal fat pad utilization, have been employed to address these issues with varying degrees of success. However, the need for predictable and stable bone regeneration and soft tissue contouring remains critical for long-term implant success.

The following study aims to assess bone gain, soft tissue contour, and stability after using bone lamina shell, providing a potential solution to enhance peri-implant tissue integrity and optimize functional and aesthetic outcomes in zygomatic implant rehabilitation.

PICOTS Population: people with atrophic maxilla. Intervention: Zygomatic implants placed in Channel shape osteotomy with using xenogenic malleable bone shell to convert osteotomy type to tunnel osteotomy.

Competitor: Zygomatic implants placed in Channel shape osteotomy with only soft tissue augmentation by using buccal bad of fat.

Outcomes:

Outcome name How to be measured Primary

Secondary • Soft tissue

* Bone gain • Measuring soft tissue thickness
* Measuring soft tissue recession.
* Measuring bone width from postoperative cone beam CT.

Time: the patient will be asked to make postoperative CT after 6 months of the surgery.

Study Design: A prospective Randomized clinical trial (two arms).

Research question:

Does the use of a xenogenic malleable bone shell in zygomatic implant rehabilitation improve bone gain, soft tissue contour and stability, thereby enhancing peri-implant tissue integrity and optimizing functional and aesthetic outcomes?"

ELIGIBILITY:
Inclusion Criteria:

1 -Patients older than 21 years. 2. Patients with severe alveolar bone atrophy in posterior maxilla (residual alveolar crest less than 5mm in height, in the area immediately distal to the canine pillar) 3. Patients with at least more than half of the zygomatic implant platform diameter inside the alveolar bone crest.

Exclusion Criteria:

1 - Patients with systemic conditions contra-indicating general anesthesia. 2. Patients with conditions contraindicating implant placement (e.g.: radiation to the head and neck, intra-venous bisphosphonates, uncontrolled Diabetes mellitus).

3. Patients with acute maxillary sinus infection or maxillary sinus cyst. 4. Restricted mouth opening (less than 3cm inter-arch distance anteriorly).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
1-soft tissue thickness 2-Soft tissue recession | 6 months of healing
  For soft tissue recession, a clinical visual exploration was performed, and defects were measured through a periodontal probe from fixed reference point (buccal surface of implant platform).
  For soft tissue thickness, a clinical method by using the average of three measurement points on the buccal side of the implant platform registered with a periodontal probe

SECONDARY OUTCOMES:
Bone gain | 6 months of healing
  CBCT used to determine bone gain in group A

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided